CLINICAL TRIAL: NCT03224169
Title: Implementation of Directly Observed Hand Hygiene in Residential Care Home for the Elderly: a Cluster Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Vincent Chi-Chung Cheng, Honorary Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QMH_MICT_1
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Multidrug Resistant Organisms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Directly observed hand hygiene
  Interventions: Behavioral: Directly observed hand hygiene
- Control (No Intervention): No directly observed hand hygiene

INTERVENTIONS:
Behavioral: Directly observed hand hygiene — Directly observed hand hygiene to the residents and staff
  Arms: Intervention

SUMMARY:
To screen the prevalence of multidrug resistant organisms among the resident in the residential care home for the elderly, and assess the practicability of directly observed hand hygiene in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Residents living the residential care home for the elderly and able to give consent

Exclusion Criteria:

* Those who cannot give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-07-18 (Estimated); Primary Completion 2017-08-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Environmental contamination | 6 weeks
  Degree of environmental contamination

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cheng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No